CLINICAL TRIAL: NCT02688764
Title: An Open-label, Randomised, Active-controlled, Parallel Group, Multicentre, Phase 3 Study to Investigate the Safety and Efficacy of PA21 (Velphoro®) and Calcium Acetate (Phoslyra®) in Paediatric and Adolescent CKD Patients With Hyperphosphataemia
Brief Title: A Study to Investigate the Safety and Efficacy of PA21 (Velphoro®) and Calcium Acetate (Phoslyra®) in Paediatric and Adolescent Chronic Kidney Disease (CKD) Patients With Hyperphosphataemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was prematurely ended due to the modification of study requirements by the US Food and Drug Administration and the European Medicines Agency
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-CL-PED-01
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Hyperphosphatemia
Keywords: PA21; phosphate binder
MeSH Terms: conditions — Hyperphosphatemia | interventions — sucroferric oxyhydroxide; calcium acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PA21 (Velphoro®) (Experimental): PA21 (Velphoro®), chewable tablets 500 mg iron
  PA21 (Velphoro®), chewable tablets 250 mg iron
  PA21 (Velphoro®), powder for oral suspension 500 mg iron
  PA21 (Velphoro®), powder for oral suspension 250 mg iron
  PA21 (Velphoro®), powder for oral suspension 125 mg iron
  Interventions: Drug: PA21 (Velphoro®)
- Calcium Acetate (Phoslyra®) (Active Comparator): Calcium Acetate (Phoslyra®) - Oral Solution: 667 mg calcium acetate per 5 mL.
  Interventions: Drug: Calcium Acetate (Phoslyra®)

INTERVENTIONS:
Drug: PA21 (Velphoro®) — During Stage 1 (Open-Label Dose Titration; up to 10 weeks), PA21 subjects will receive PA21 at a starting dose based on their age. Dose of PA21 will be increased or decreased as required for efficacy (to achieve age specific target serum phosphorus level), provided a subject has been receiving that dose for a minimum of 2 weeks, and for safety or tolerability reasons at any time.
  During Stage 2 (Open-Label Safety Extension, 24 week safety extension),subjects will continue on the dose received at the end of Stage 1, unless a dose change is required. Doses may be titrated for efficacy (to achieve age specific target Serum phosphorus levels), provided a subject has been receiving that dose for a minimum of 2 weeks, and for safety or tolerability reasons at any time during Stage 2.
  Other Names: sucroferric oxyhydroxide
  Arms: PA21 (Velphoro®)
Drug: Calcium Acetate (Phoslyra®) — During Stage 1 (Open-Label Dose Titration; up to 10 weeks), Phoslyra subjects will receive Phoslyra either at a starting dose based on their weight or, if considered more appropriate by the Investigator, at an equivalent dose of their previous phosphate binder (PB), calcium-based or sevelamer. Dose of Phoslyra will be increased or decreased as required for efficacy (to achieve age specific target serum phosphorus level), provided a subject has been receiving that dose for a minimum of 2 weeks, and for safety or tolerability reasons at any time.
  During Stage 2 (Open-Label Safety Extension, 24 week safety extension),subjects will continue on the dose received at the end of Stage 1, unless a dose change is required. Doses may be titrated for efficacy (to achieve age specific target Serum phosphorus levels), provided a subject has been receiving that dose for a minimum of 2 weeks, and for safety or tolerability reasons at any time during Stage 2.
  Arms: Calcium Acetate (Phoslyra®)

SUMMARY:
This is a Phase 3, Open-label, Randomised, Active-controlled, Parallel Group, Multicentre Study to Investigate the Safety and Efficacy of PA21 (Velphoro®) and Calcium Acetate (Phoslyra®) in Paediatric and Adolescent CKD Patients with Hyperphosphataemia. The aim of this Phase 3 clinical study is to demonstrate similar efficacy of PA21 (Velphoro) in paediatric and adolescent patients with CKD, and to provide safety and dosing information for this patient population. The Phoslyra (comparator) group provides information for a descriptive comparison of PA21 against a commonly used calcium-based phosphate binder (calcium acetate).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 0 to <18 years at time of consent.
2. Subjects with hyperphosphataemia
3. Subjects ≥1 year with CKD Stages 4-5 defined by a glomerular filtration rate <30 mL/min/1.73 m2 or with CKD Stage 5D receiving adequate maintenance haemodialysis (HD) or peritoneal dialysis (PD) for at least 2 months prior to screening.
4. Subjects <1 year must have CKD.
5. Appropriate written informed consent and, where appropriate/required assent, have been provided.

Exclusion Criteria:

1. Subjects with hypercalcaemia at screening
2. Subjects with intact parathyroid hormone (iPTH) levels >700 pg/mL at screening.
3. Subjects who are PB naïve who weigh <5 kg at screening. Subjects receiving stable doses of PBs who weigh <6 kg at screening
4. Subjects requiring feeding tube sizes ≤6 FR (French catheter scale).
5. Subjects with history of major gastrointestinal surgery or significant gastrointestinal disorders.
6. Subjects with hypocalcaemia (serum total corrected calcium <1.9 mmol/L; <7.6 mg/dL) at screening.
7. Subject is pregnant (e.g., positive human chorionic gonadotropin test) or breast feeding.
8. Subject has a significant medical condition(s)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Greenbaum, MD; PhD, Principal Investigator — Children's Healthcare of Atlanta at Egleston
Locations (38):
- United States (22):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Emory-Children's Center, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - The University of New Mexico, Albuquerque, New Mexico
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Doernbecher Children's Hospital, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital - Texas Children's Feigin Center, Houston, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - Hôpital Jeanne de Flandre, Lille
  - Chu de Lyon - Hopital Femme Mere Enfant, Lyon
  - Service de Néphrologie et Endocrinologie pédiatriques, Montpellier
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
- Lithuania (2):
  - Hospital Of Lithuanian University Of Health Sciences Kaunas Clinics, Kaunas
  - Children's Hospital, Affiliate of Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Poland (4):
  - Uniwersytecki Dziecięcy Szpital Kliniczny im. L. Zamenhofa w Białymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie - Prokocimiu, Krakow
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
- Romania (2):
  - Spitalul Clinic de Urgenţă pentru copii "Maria Sklodowska Curie", Bucharest, Bucharest
  - Spitalul Clinic Fundeni Bucureşti, Bucharest, Bucharest
- Russia (3):
  - Children's Republican Clinical Hospital, Kazan'
  - St. Vladimir Children's City Clinical Hospital, Moscow
  - St. Petersburg GBUZ "Children's City Hospital No. 1", Saint Petersburg

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- PA21 (Velphoro®): Formulations:
  PA21 (Velphoro®), chewable tablets 500 mg and 250 mg iron
  PA21 (Velphoro®), powder for oral suspension 500 mg, 250 mg and 125 mg iron
  Stage 1 (Open-Label Dose Titration; up to 10 weeks): starting dose based on the participant's age. Dose was increased or decreased as required for efficacy (to achieve age specific target serum phosphorus level), provided a subject had been receiving that dose for a minimum of 2 weeks, and for safety/tolerability reasons at any time.
  Stage 2 (Open-Label Safety Extension, 24 week safety extension): dose received at the end of Stage 1, unless a dose change is required. Doses could be titrated for efficacy (to achieve age specific target Serum phosphorus levels), provided a subject had been receiving that dose for a minimum of 2 weeks, and for safety or tolerability reasons at any time.
- Calcium Acetate (Phoslyra®): Formulation:
  Calcium Acetate (Phoslyra®) - Oral Solution: 667 mg calcium acetate per 5 mL.
  Stage 1 (Open-Label Dose Titration; up to 10 weeks): starting dose based on the participant's weight or, if considered more appropriate by the Investigator, at an equivalent dose of their previous phosphate binder (PB), calcium-based or sevelamer. Dose was increased or decreased as required for efficacy (to achieve age specific target serum phosphorus level), provided a subject had been receiving that dose for a minimum of 2 weeks, and for safety/tolerability reasons at any time.
  Stage 2 (Open-Label Safety Extension, 24 week safety extension): dose received at the end of Stage 1, unless a dose change is required. Doses could be titrated for efficacy (to achieve age specific target Serum phosphorus levels), provided a subject had been receiving that dose for a minimum of 2 weeks, and for safety/tolerability reasons at any time.
Period: Overall Study
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Started | 66 | 19
Treated in Stage 1 | 66 | 19
Treated in Stage 2 | 43 | 8
Completed | 26 | 2
Not Completed | 40 | 17
Not completed — Adverse Event | 3 | 3
Not completed — AE/Kidney transplant | 1 | 0
Not completed — AE/Lack of efficacy | 1 | 0
Not completed — AE/Non-compl. | 1 | 0
Not completed — AE/Non-compl./Withd. parent | 0 | 1
Not completed — AE/Other | 0 | 1
Not completed — AE/Physician decision | 1 | 0
Not completed — AE/Withd. parent | 3 | 0
Not completed — AE/Withd. parent/Withd. subject | 1 | 1
Not completed — AE/Withd. subject | 1 | 0
Not completed — Kidney transplant | 10 | 4
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lack of efficacy/Physician decision | 0 | 1
Not completed — Non-compliance with study drug | 4 | 0
Not completed — Non-compl./Physician decision | 2 | 0
Not completed — Non-compl./Ph. decision/Withd. subject | 1 | 1
Not completed — Non-compl./Withd. subject | 0 | 2
Not completed — Phosphorus level outside safe range | 0 | 1
Not completed — Phosphorus >7 mg/dL - Withd. by sponsor | 1 | 0
Not completed — Study drug taste/Withd. parent | 1 | 0
Not completed — Subject moving out | 2 | 0
Not completed — Subject taken off dialysis | 1 | 0
Not completed — Withdrawal by parent | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®) | Total
Number analyzed (Participants) | 66 | 19 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (4.07) | 12.6 (3.73) | 12.3 (3.98)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: Newborns (0-27 days) | 0 | 0 | 0
  Age, Categorical: Infants (28 days-23 months) | 0 | 0 | 0
  Age, Categorical: Children (2-11 years) | 23 | 6 | 29
  Age, Categorical: Adolescents (12-17 years) | 42 | 13 | 55
  Age, Categorical: Adults (18-64 years) | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 13 | 47
  Male | 32 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 5 | 25
  Not Hispanic or Latino | 46 | 14 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 9 | 2 | 11
  White | 43 | 14 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 39 | 14 | 53
  France | 6 | 0 | 6
  Lithuania | 3 | 0 | 3
  Poland | 4 | 2 | 6
  Germany | 5 | 1 | 6
  Russia | 1 | 1 | 2
  Romania | 8 | 1 | 9
Height [Mean (Standard Deviation); unit: cm] | 142.3 (24.10) | 140.3 (24.12) | 141.9 (23.98)
Weight [Mean (Standard Deviation); unit: kg] | 41.90 (18.023) | 38.28 (17.834) | 41.10 (17.939)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 19.621 (4.6182) | 18.483 (4.4238) | 19.366 (4.5743)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphorus Level From Baseline to the End of Stage 1 in the PA21 Group
Time Frame: From Baseline to the End of Stage 1 (up to 10 weeks after treatment start date)
Population: Full Analysis Set (FAS) Population: all participants randomised to treatment at Stage 1 who received at least 1 dose of randomised treatment and who had at least 1 post-baseline assessment of the efficacy endpoint (serum phosphorus level), analysed according to treatment randomised.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- PA21 (Velphoro®): Formulations:
  PA21 (Velphoro®), chewable tablets 500 mg and 250 mg iron PA21 (Velphoro®), powder for oral suspension 500 mg, 250 mg and 125 mg iron
  Stage 1 (Open-Label Dose Titration; up to 10 weeks): starting dose based on the participant's age. Dose was increased or decreased as required for efficacy (to achieve age specific target serum phosphorus level), provided a subject had been receiving that dose for a minimum of 2 weeks, and for safety/tolerability reasons at any time.
Arm/Group | PA21 (Velphoro®)
Number analyzed (Participants) | 65
mmol/L | -0.120 (0.081)
Statistical Analysis 1: Comparison: PA21 (Velphoro®); Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 1 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.1465, t-test, 2 sided — 0.05 level of significance

2. Primary Outcome: Number and Percentage of Participants Who Withdrew Due to Treatment Emergent Adverse Events
Description: Any adverse event Leading to Study Drug Withdrawal is considered.
Time Frame: through study completion, up to 34 weeks after treatment start date
Population: Safety Population: all participants who received at least 1 dose of study medication, analysed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
Participants | 12 | 6

3. Primary Outcome: Number and Percentage of Participants With Any Treatment Emergent Adverse Event
Description: Please note that in this section we are presenting just the overview of the adverse events experienced by the trial participants, in particular, the number of participants with at least one TEAEs until end of stage 2.
  Please refer to the detailed tables included on the Adverse Event Module for specifics.
Time Frame: through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
Participants | 50 | 14

4. Secondary Outcome: Change in Serum Phosphorus Level From Baseline to the End of Stage 1 in the Phoslyra Group
Time Frame: From Baseline to the End of Stage 1 (up to 10 weeks after treatment start date)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- Calcium Acetate (Phoslyra®): Formulation:
  Calcium Acetate (Phoslyra®) - Oral Solution: 667 mg calcium acetate per 5 mL.
  Stage 1 (Open-Label Dose Titration; up to 10 weeks): starting dose based on the participant's weight or, if considered more appropriate by the Investigator, at an equivalent dose of their previous phosphate binder (PB), calcium-based or sevelamer. Dose was increased or decreased as required for efficacy (to achieve age specific target serum phosphorus level), provided a subject had been receiving that dose for a minimum of 2 weeks, and for safety/tolerability reasons at any time.
Arm/Group | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 15
mmol/L | -0.615 (0.320)
Statistical Analysis 1: Comparison: Calcium Acetate (Phoslyra®); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0872, t-test, 2 sided — 0.05 level of significance

5. Secondary Outcome: Change in Serum Phosphorus Level From Baseline to the End of Stage 2 in Both Groups
Time Frame: From baseline to study completion, up to 34 weeks after treatment start date
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 36 | 6
mmol/L | 0.099 (0.198) | -0.393 (0.218)
Statistical Analysis 1: Comparison: PA21 (Velphoro®); Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 2 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.6207, t-test, 2 sided — 0.05 level of significance
Statistical Analysis 2: Comparison: Calcium Acetate (Phoslyra®); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.3226, t-test, 2 sided — 0.05 level of significance

6. Secondary Outcome: Participants With Serum Phosphorus Levels Within the Age-dependent Target Range in Each Stage
Description: Number and percentages of participants with serum phosphorus levels below, within and above age-dependent target ranges at baseline, at the end of Stage 1 and at the end of Stage 2.
  The age target ranges for serum phosphorus levels are:
  * 0 to <1 year 1.62-2.52 mmol/L
  * 1 year to <6 years 1.45-2.10 mmol/L
  * 6 years to <13 years 1.16-1.87 mmol/L
  * 13 years to ≤18 years 0.74-1.45 mmol/L
Time Frame: through study completion, up to 34 weeks after treatment start date
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 65 | 15
Participants
  Baseline: Below | 2 | 1
  Baseline: Within | 11 | 1
  Baseline: Above | 52 | 13
  End of Stage 1: number analyzed (Participants) | 64 | 15
  End of Stage 1: Below | 2 | 1
  End of Stage 1: Within | 25 | 2
  End of Stage 1: Above | 37 | 12
  End of Stage 2: number analyzed (Participants) | 40 | 8
  End of Stage 2: Below | 1 | 0
  End of Stage 2: Within | 14 | 2
  End of Stage 2: Above | 25 | 6

7. Secondary Outcome: Participants With Serum Phosphorus Levels Within the Age Related Normal Range in Each Stage
Description: Number and percentages of participants with serum phosphorus levels below, within and above age-dependent normal ranges at baseline, at the end of Stage 1 and at the end of Stage 2.
  The age related normal ranges for serum phosphorus levels are:
  * 0 to <1year 1.36 - 2.62 mmol/L
  * 1 year to <6 years 1.03 - 1.97 mmol/L
  * 6 years to <9 years 1.03 - 1.97 mmol/L
  * 9 years to <10 years 1.03 - 1.97 mmol/L
  * 10 years to <15 years 1.00 - 1.94 mmol/L
  * 15 years to ≤18 years 0.71 - 1.65 mmol/L
Time Frame: through study completion, up to 34 weeks after treatment start date
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 65 | 15
Participants
  Baseline: Below | 1 | 1
  Baseline: Within | 24 | 5
  Baseline: Above | 40 | 9
  End of Stage 1: number analyzed (Participants) | 64 | 15
  End of Stage 1: Below | 1 | 1
  End of Stage 1: Within | 39 | 6
  End of Stage 1: Above | 24 | 8
  End of Stage 2: number analyzed (Participants) | 40 | 8
  End of Stage 2: Below | 1 | 0
  End of Stage 2: Within | 23 | 2
  End of Stage 2: Above | 16 | 6

8. Secondary Outcome: Serum Phosphorus Values at Each Visit
Time Frame: through study completion, up to 34 weeks after treatment start date
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 65 | 15
mmol/L
  Baseline | 2.07 (0.522) | 2.15 (0.669)
  End of Stage 1: number analyzed (Participants) | 64 | 15
  End of Stage 1 | 1.82 (0.575) | 2.17 (0.804)
  End of Stage 2: number analyzed (Participants) | 40 | 8
  End of Stage 2 | 1.71 (0.506) | 2.09 (0.594)

9. Secondary Outcome: Serum Total Corrected Calcium at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
mmol/L
  Baseline | 2.38 (0.144) | 2.37 (0.185)
  End of Stage 1 - Observed data: number analyzed (Participants) | 65 | 17
  End of Stage 1 - Observed data | 2.35 (0.212) | 2.31 (0.130)
  End of Stage 2 - Observed data: number analyzed (Participants) | 41 | 8
  End of Stage 2 - Observed data | 2.28 (0.185) | 2.36 (0.154)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 65 | 17
  End of Stage 1 - Change from baseline | -0.03 (0.224) | -0.06 (0.212)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 41 | 8
  End of Stage 2 - Change from baseline | -0.06 (0.197) | -0.07 (0.207)

10. Secondary Outcome: Participants With Sustained Hypercalcaemia
Description: Number and percentages of participants with at least 1 episode of sustained hypercalcaemia (defined as total calcium value above the upper safety limit confirmed by repeat sample 1 week later) during the study
Time Frame: through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
Participants | 6 | 4

11. Secondary Outcome: Serum Total Corrected Calcium-Phosphorus Product at Each Time Point and Change From Baseline
Description: Summary statistics of Serum total corrected calcium-phosphorus product at each time point and change from baseline, where serum total corrected calcium-phosphorus product correspond to the product of serum total calcium and Phosphorus, expressed in mmol^2/L^2
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol^2/L^2
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
mmol^2/L^2
  Baseline | 4.94 (1.400) | 5.31 (1.831)
  End of Stage 1 - Observed data: number analyzed (Participants) | 65 | 17
  End of Stage 1 - Observed data | 4.25 (1.392) | 5.05 (1.608)
  End of Stage 2 - Observed data: number analyzed (Participants) | 40 | 8
  End of Stage 2 - Observed data | 3.91 (1.211) | 4.90 (1.289)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 65 | 17
  End of Stage 1 - Change from baseline | -0.65 (1.221) | -0.31 (2.152)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 40 | 8
  End of Stage 2 - Change from baseline | -0.49 (1.384) | -0.12 (1.227)

12. Secondary Outcome: Serum iPTH Levels at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
pmol/L
  Baseline: number analyzed (Participants) | 65 | 19
  Baseline | 30.36 (26.393) | 37.12 (19.527)
  End of Stage 1 - Observed data: number analyzed (Participants) | 64 | 15
  End of Stage 1 - Observed data | 28.28 (20.972) | 45.90 (28.363)
  End of Stage 2 - Observed data: number analyzed (Participants) | 41 | 8
  End of Stage 2 - Observed data | 35.60 (32.903) | 52.30 (36.143)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 64 | 15
  End of Stage 1 - Change from baseline | -2.49 (22.139) | 5.72 (20.166)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 40 | 8
  End of Stage 2 - Change from baseline | 4.61 (38.858) | 12.01 (27.151)

13. Secondary Outcome: Ferritin Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
ug/L
  Baseline: number analyzed (Participants) | 56 | 16
  Baseline | 223.67 (274.071) | 234.28 (228.825)
  End of Stage 1 - Observed data: number analyzed (Participants) | 58 | 15
  End of Stage 1 - Observed data | 322.59 (368.823) | 310.46 (369.869)
  End of Stage 2 - Observed data: number analyzed (Participants) | 33 | 8
  End of Stage 2 - Observed data | 326.13 (304.864) | 345.13 (366.230)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 51 | 14
  End of Stage 1 - Change from baseline | 48.59 (168.999) | 59.27 (219.660)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 28 | 8
  End of Stage 2 - Change from baseline | 137.57 (149.176) | 110.69 (211.054)

14. Secondary Outcome: Unsaturated Iron Binding Capacity Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
umol/L
  Baseline: number analyzed (Participants) | 65 | 19
  Baseline | 28.68 (12.985) | 25.54 (14.153)
  End of Stage 1 - Observed data: number analyzed (Participants) | 64 | 16
  End of Stage 1 - Observed data | 25.37 (11.162) | 27.28 (9.671)
  End of Stage 2 - Observed data: number analyzed (Participants) | 40 | 8
  End of Stage 2 - Observed data | 25.53 (11.672) | 26.04 (11.088)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 63 | 16
  End of Stage 1 - Change from baseline | -3.64 (9.284) | -0.81 (7.176)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 39 | 8
  End of Stage 2 - Change from baseline | -4.38 (12.454) | -3.53 (11.779)

15. Secondary Outcome: Iron Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
umol/L
  Baseline: number analyzed (Participants) | 65 | 19
  Baseline | 13.20 (6.948) | 15.25 (8.488)
  End of Stage 1 - Observed data: number analyzed (Participants) | 64 | 16
  End of Stage 1 - Observed data | 14.70 (7.425) | 12.66 (4.821)
  End of Stage 2 - Observed data: number analyzed (Participants) | 40 | 8
  End of Stage 2 - Observed data | 14.31 (6.005) | 13.08 (4.967)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 63 | 16
  End of Stage 1 - Change from baseline | 1.64 (8.946) | -0.18 (7.197)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 39 | 8
  End of Stage 2 - Change from baseline | 1.95 (6.940) | 1.35 (9.691)

16. Secondary Outcome: Transferrin Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
g/L
  Baseline | 2.12 (0.607) | 1.99 (0.565)
  End of Stage 1 - Observed data: number analyzed (Participants) | 65 | 16
  End of Stage 1 - Observed data | 1.96 (0.520) | 1.97 (0.588)
  End of Stage 2 - Observed data: number analyzed (Participants) | 41 | 8
  End of Stage 2 - Observed data | 1.89 (0.513) | 1.98 (0.439)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 65 | 16
  End of Stage 1 - Change from baseline | -0.17 (0.342) | -0.05 (0.234)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 41 | 8
  End of Stage 2 - Change from baseline | -0.28 (0.506) | -0.12 (0.289)

17. Secondary Outcome: 25-Hydroxy Vitamin D Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
nmol/L
  Baseline: number analyzed (Participants) | 56 | 17
  Baseline | 83.1 (38.74) | 81.7 (40.32)
  End of Stage 1 - Observed data: number analyzed (Participants) | 31 | 10
  End of Stage 1 - Observed data | 79.8 (34.25) | 74.4 (38.68)
  End of Stage 2 - Observed data: number analyzed (Participants) | 32 | 8
  End of Stage 2 - Observed data | 76.0 (37.48) | 59.0 (17.18)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 26 | 10
  End of Stage 1 - Change from baseline | -4.1 (24.28) | -9.7 (22.68)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 27 | 8
  End of Stage 2 - Change from baseline | -18.3 (27.77) | -21.8 (15.28)

18. Secondary Outcome: Bone Specific Alkaline Phosphatase Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
ug/L
  Baseline: number analyzed (Participants) | 55 | 17
  Baseline | 47.77 (35.469) | 55.55 (50.249)
  End of Stage 1 - Observed data: number analyzed (Participants) | 31 | 10
  End of Stage 1 - Observed data | 50.37 (42.382) | 56.15 (64.537)
  End of Stage 2 - Observed data: number analyzed (Participants) | 32 | 8
  End of Stage 2 - Observed data | 55.31 (43.363) | 71.46 (64.427)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 26 | 10
  End of Stage 1 - Change from baseline | 7.29 (28.837) | 2.38 (27.375)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 26 | 8
  End of Stage 2 - Change from baseline | 7.74 (41.156) | -4.18 (38.713)

19. Secondary Outcome: Type I Collagen C-Telopeptides Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
ug/L
  Baseline: number analyzed (Participants) | 54 | 17
  Baseline | 4.77 (1.201) | 4.31 (1.549)
  End of Stage 1 - Observed data: number analyzed (Participants) | 32 | 9
  End of Stage 1 - Observed data | 4.57 (1.549) | 5.10 (1.799)
  End of Stage 2 - Observed data: number analyzed (Participants) | 29 | 7
  End of Stage 2 - Observed data | 4.21 (1.591) | 4.43 (1.565)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 26 | 9
  End of Stage 1 - Change from baseline | -0.45 (1.387) | -0.03 (1.217)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 23 | 7
  End of Stage 2 - Change from baseline | -0.42 (1.893) | -0.34 (0.970)

20. Secondary Outcome: Fibroblast Growth Factor 23 Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
pg/mL
  Baseline: number analyzed (Participants) | 53 | 14
  Baseline | 820.1 (503.90) | 814.9 (468.89)
  End of Stage 1 - Observed data: number analyzed (Participants) | 29 | 8
  End of Stage 1 - Observed data | 775.7 (514.86) | 767.7 (482.47)
  End of Stage 2 - Observed data: number analyzed (Participants) | 32 | 6
  End of Stage 2 - Observed data | 603.5 (531.86) | 747.4 (628.27)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 23 | 7
  End of Stage 1 - Change from baseline | -60.7 (454.95) | -41.8 (729.27)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 27 | 5
  End of Stage 2 - Change from baseline | -187.6 (507.26) | 47.8 (467.87)

21. Secondary Outcome: Osteocalcin-CL Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
ug/L
  Baseline: number analyzed (Participants) | 54 | 17
  Baseline | 517.9 (357.11) | 681.5 (445.94)
  End of Stage 1 - Observed data: number analyzed (Participants) | 29 | 9
  End of Stage 1 - Observed data | 586.0 (421.72) | 753.1 (412.38)
  End of Stage 2 - Observed data: number analyzed (Participants) | 32 | 8
  End of Stage 2 - Observed data | 516.9 (429.24) | 709.0 (462.59)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 23 | 9
  End of Stage 1 - Change from baseline | 28.4 (248.44) | 20.0 (179.26)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 27 | 8
  End of Stage 2 - Change from baseline | 20.3 (342.77) | -91.0 (200.09)

22. Secondary Outcome: Tartrate-resistant Acid Phosphatase 5b Values at Each Time Point and Change From Baseline
Time Frame: From baseline through study completion, up to 34 weeks after treatment start date
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
Number analyzed (Participants) | 66 | 19
U/L
  Baseline: number analyzed (Participants) | 50 | 15
  Baseline | 8.86 (7.646) | 8.82 (5.161)
  End of Stage 1 - Observed data: number analyzed (Participants) | 30 | 9
  End of Stage 1 - Observed data | 8.55 (8.305) | 8.82 (5.160)
  End of Stage 2 - Observed data: number analyzed (Participants) | 29 | 5
  End of Stage 2 - Observed data | 8.25 (5.643) | 7.62 (2.044)
  End of Stage 1 - Change from baseline: number analyzed (Participants) | 23 | 8
  End of Stage 1 - Change from baseline | 0.02 (2.746) | -0.11 (4.580)
  End of Stage 2 - Change from baseline: number analyzed (Participants) | 23 | 5
  End of Stage 2 - Change from baseline | 0.72 (4.108) | -0.16 (2.422)

23. Post Hoc Outcome: Change in Serum Phosphorus Level From Baseline to End of Stage 1 in PA21 Group, by Age Group
Time Frame: From Baseline to the End of Stage 1 (up to 10 weeks after treatment start date)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PA21 (Velphoro®)
Number analyzed (Participants) | 65
mmol/L
  <2 years: number analyzed (Participants) | 0
  >=2 years to <6 years: number analyzed (Participants) | 6
  >=2 years to <6 years | -0.078 (0.123)
  >=6 years to <12 years: number analyzed (Participants) | 17
  >=6 years to <12 years | -0.200 (0.158)
  >=12 years to <=18 years: number analyzed (Participants) | 42
  >=12 years to <=18 years | -0.149 (0.062)
Statistical Analysis 1: Comparison: PA21 (Velphoro®); Age group of >=2 years to <6 years Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 1 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.5682, t-test, 2 sided — 0.05 level of significance
Statistical Analysis 2: Comparison: PA21 (Velphoro®); Age group of >=6 years to <12 years Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 1 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.2271, t-test, 2 sided — 0.05 level of significance
Statistical Analysis 3: Comparison: PA21 (Velphoro®); Age group of >=12 years to <=18 years Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 1 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.0220, t-test, 2 sided — 0.05 level of significance

24. Post Hoc Outcome: Change in Serum Phosphorus (SP) Level From Baseline to End of Stage 1 in PA21 Group, by Serum Phosphorus Level at Baseline
Description: The levels of Serum Phosphorus considered at baseline are those above vs within/below Age Related Normal Range
Time Frame: From Baseline to the End of Stage 1 (up to 10 weeks after treatment start date)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PA21 (Velphoro®)
Number analyzed (Participants) | 65
mmol/L
  SP above Age Related Normal Range: number analyzed (Participants) | 40
  SP above Age Related Normal Range | -0.282 (0.096)
  SP below/within Related Normal Range: number analyzed (Participants) | 25
  SP below/within Related Normal Range | 0.082 (0.146)
Statistical Analysis 1: Comparison: PA21 (Velphoro®); Group of SP at baseline above Age Related Normal Range Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 1 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.0058, t-test, 2 sided — 0.05 level of significance
Statistical Analysis 2: Comparison: PA21 (Velphoro®); Group of SP at baseline below or within Age Related Normal Range Results are obtained from a linear mixed model which includes change in serum phosphorus levels from baseline to the end of Stage 1 as dependent variable and treatment, baseline serum phosphorus, age (in categories) at randomisation, region (Non-US/US) and gender as fixed effects; Test type: Superiority; p = 0.5801, t-test, 2 sided — 0.05 level of significance

ADVERSE EVENTS:
Time Frame: Through study completion, up to 34 weeks after treatment start date
Description: TEAEs (treatment emergent adverse events) are included in this section.
Arm/Group | PA21 (Velphoro®) | Calcium Acetate (Phoslyra®)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/19
Serious Adverse Events (participants affected / at risk) | 18/66 | 3/19
Other Adverse Events (participants affected / at risk) | 45/66 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA21 (Velphoro®) (N=66) | Calcium Acetate (Phoslyra®) (N=19)
Weight increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (6) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Puncture site reaction (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 2 (3) | 0 (0)
Device extrusion (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0)
Benign intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA21 (Velphoro®) (N=66) | Calcium Acetate (Phoslyra®) (N=19)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperparathyroidism (Endocrine disorders) | 2 (3) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (2) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely ended as a result of the modification of study requirements, as agreed with the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results of the Services or other information on the Clinical Study may be disclosed or submitted for publication or presentation without the Sponsor's prior written agreement.

DOCUMENTS (2):
  • Study Protocol (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02688764/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT02688764/SAP_001.pdf